CLINICAL TRIAL: NCT02098876
Title: Evaluation of WSS and Neointimal Healing Following Percutaneous Coronary Intervention of Angulated Vessels With Resolute® Integrity Zotarolimus Eluting Coronary Stent Compared to XIENCE Xpedition® Everolimus Eluting Coronary Stent
Brief Title: Wall Shear Stress and Neointimal Healing Following PCI in Angulated Coronary Vessels
Acronym: SHEAR-STENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Habib Samady, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00066353
Record Dates: First submitted 2014-01-10; First posted 2014-03-28 (Estimated); Results first posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-08

CONDITIONS: Coronary Artery Disease
Keywords: neointimal tissue area; angulated coronary vessels; wall shear stress; zotarolimus eluting stent; everolimus eluting stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Tomography, Optical Coherence; Ultrasonography, Interventional

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Resolute Integrity DES (Active Comparator): Resolute Integrity zotarolimus eluting stent
  Interventions: Device: Resolute Integrity Zotarolimus eluting stent; Device: Optical Coherence Tomography (OCT); Device: Intravascular Ultrasound (IVUS)
- Xience Xpedition DES (Active Comparator): Xience Xpedition everolimus eluting stent
  Interventions: Device: Xience Xpedition everolimus eluting stent; Device: Optical Coherence Tomography (OCT); Device: Intravascular Ultrasound (IVUS)

INTERVENTIONS:
Device: Resolute Integrity Zotarolimus eluting stent — PCI with Resolute stent
  Arms: Resolute Integrity DES
Device: Xience Xpedition everolimus eluting stent — PCI with Xience stent
  Arms: Xience Xpedition DES
Device: Optical Coherence Tomography (OCT) — Optical coherence tomography (OCT) will be performed at baseline to assess plaque burden prior to and after stent deployment as well as to evaluate stent expansion and stent apposition. OCT will be repeated at one year follow-up to evaluate neo-intimal tissue coverage within the stent and change in plaque area at the stent edges. Offline, manual detection of lumen area and stent area will be performed for each OCT cross-section from baseline and follow up examinations.
Device: Intravascular Ultrasound (IVUS) — Intravascular ultrasound (IVUS) will be performed at baseline to assess plaque burden prior to and after stent deployment as well as to evaluate stent expansion and stent apposition. IVUS will be repeated at one year follow-up to evaluate neo-intimal tissue coverage within the stent and change in plaque area at the stent edges. Offline, manual detection of lumen area, stent area, vessel area (external elastic membrane) and the media-adventitia interface will be performed for each IVUS cross-section from baseline and follow up examinations.

SUMMARY:
Stents are metallic tubular supports placed inside a blood vessel to relieve an obstruction and restore blood flow to the heart muscle. Stents could also be coated with a drug (drug-eluting stents - DES) that improves local healing and inhibits growth of scar tissue within the vessel that otherwise could lead to re-narrowing. This study will evaluate the effects of 2 FDA-approved metallic stents with different designs that may have important effects on regional plaque response and blood flow dynamics immediately after stent deployment and stent healing at 12 months follow up.

DETAILED DESCRIPTION:
The past two decades have registered major advances in cardiovascular medicine that have improved patients' survival and quality of life. One area of major research and innovation is the field of percutaneous coronary interventions (PCI), a non-surgical procedure used to treat a narrowed heart artery with stents. Stents are metallic tubular supports placed inside a blood vessel to relieve an obstruction and restore blood flow to the heart muscle. Stents could also be coated with a drug (drug-eluting stents - DES) that improves local healing and inhibits growth of scar tissue (smooth muscle and fibrous cells) within the vessel that otherwise could lead to re-narrowing.

The investigators study will evaluate two FDA-approved DES, currently in use, with respect to coronary vessel healing and long term patency. These include the XIENCE Xpedition Everolimus drug-eluting stent (X-EES) from Abbott Vascular and Resolute Integrity® Zotarolimus drug-eluting stent (R-ZES) from Medtronic, Inc, both of which have been shown in large clinical trials to be safe and effective. This study will evaluate the effects of apparently subtle differences in stent design between these two platforms that may have important effects on regional plaque response and blood flow dynamics immediately after stent deployment and stent healing and scar formation at 12 months follow up.

Several aspect of the R-ZES compared to the X-EES design may result in more favorable regional plaque response and blood flow dynamics immediately after stent deployment. These include a more compliant stent design made of a single sinusoidal wire with no connector between struts that is likely to be more comformable to a curved or angulated coronary vessels. In heart vessels which are not angulated, these features may not make a major difference in outcomes as studies already suggest. Whereas, in narrowed arteries which are curved or angulated, the use of X-EES could result in more straightening of the vessel's natural curvature and more disturbance in flow patterns. In contrast, the use of R-ZES in angulated arteries could cause less hemodynamic disturbances. There is a great deal of data suggesting that disturbances in local blood flow patterns and creation of eddy currents ('turbulent' blood flow) could adversely affect stent healing and exacerbate neointimal tissue growth.

Using two intravascular imaging technologies, the optical coherence tomography (OCT) and intravascular ultrasound (IVUS), this study aims to investigate differences in scar tissue coverage within the stented region and the degree of narrowing at the edges of the stent in patients undergoing clinically-indicated PCI (with R-ZES and X-EES) at 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be 30 to 80 years old
2. Severe coronary lesion in a vessel with ≥ 30-degree angulation requiring percutaneous coronary intervention (PCI)
3. Lesion treatable by a single Resolute Integrity or Onyx Abbott Xience Xpedition or Sierra coronary drug-eluting stent.
4. Patients with stable ischemic heart disease or acute coronary syndrome undergoing clinically PCI.

Exclusion Criteria:

1. Inability to provide informed consent prior to randomization
2. Anatomy requiring coronary artery bypass surgery (CABG)
3. History of prior CABG in the territory of the vessel being considered for PCI
4. Heavily calcified lesion requiring rotablation or other debulking or scoring device for successful stent deployment
5. Large thrombus burden on recent angiography
6. Previously stented vessels
7. Ostial lesions: lesion located within 5mm of the origin of the left anterior descending artery (LAD), left circumflex artery (LCx), or Right coronary artery (RCA)
8. Lesions at bifurcations and those that occlude side branches >2.5mm
9. Recent (<72 hours) ST-elevation myocardial infarction (STEMI).
10. Planned surgical procedures in the subsequent 12 months
11. History of hypersensitivity or contraindication to device materials and their degradants, everolimus, zotarolimus, cobalt, chromium, nickel, platinum, tungsten, acrylic, and fluoropolymers
12. History of any solid organ transplantation or subject is on a waiting list for any solid organ transplant
13. Left ventricular ejection fraction < 30%
14. Known allergies to clinically utilized anti-thrombotic or anti-platelet agents
15. Unable to tolerate long term dual antiplatelet therapy
16. Pregnancy or lactation

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Habib Samady, MD, Principal Investigator — Georgia Heart Institute, Northeast Georgia Medical Center
Locations (10):
- Emory University, Atlanta, Georgia, United States
- Nanjing Medical University, Nanjing Heart Center, Nanjing, China
- Japan (2):
  - Kobe University Graduate School of Medicine, Hyōgo
  - Wakayama Medical University Department of Cardiovascular Medicine, Wakayama
- Latvian Society of Cardiology Pauls Stradins Clinical University Hospital, Riga, Latvia
- University Clinical Center of Serbia, Belgrade, Serbia
- South Korea (3):
  - Seoul National University College of Medicine, Seoul
  - Samsung Medical Center, Sungkyunkwan University School of Medicine Division of Cardiology, Seoul
  - Ulsan University Hospital University of Ulsan College of Medicine, Ulsan
- Hospital Clinico San Carlos, Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Molony DS, Hung O, Corban M, Gogas B, Lefieux A, Shah I, Komilian K, Adams A, Sykalo C, Dodoo S, Kumar A, Kumar S, Azarnoosh J, Piccinelli M, McDaniel MC, King SB, Maynard C, Chatzizisis YS, Chen SL, Shin ES, Stankovic G, Milasinovic D, Erglis A, Otake H, Akasaka T, Escaned J, Kwon-Koo B, Wook-Nam C, Won KB, Murasato Y, Lee WY, Lee SH, Hahn JY, Lee JM, Giddens DP, Veneziani A, Samady H. A randomized prospective study investigating the relationship between post-PCI wall shear stress and 12-month neointimal healing: The SHEAR-STENT study. Cardiovasc Revasc Med. 2025 Nov 15:S1553-8389(25)00569-X. doi: 10.1016/j.carrev.2025.11.001. Online ahead of print. PMID 41285658

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 12 SITES. Participant enrollment began in May 2014 and all follow up was complete by December 2020.
Period: Overall Study
Arm/Group | Resolute Integrity DES | Xience Xpedition DES
Started | 45 | 41
Completed | 40 | 36
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resolute Integrity DES | Xience Xpedition DES | Total
Number analyzed (Participants) | 45 | 41 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 23 | 49
  >=65 years | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (11.6) | 63.8 (10.6) | 63.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 36 | 34 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 30 | 31 | 61
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 12 | 8 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  South Korea | 13 | 13 | 26
  Latvia | 1 | 0 | 1
  United States | 6 | 4 | 10
  China | 9 | 6 | 15
  Japan | 8 | 12 | 20
  Serbia | 7 | 6 | 13
  Spain | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: In Stent Mean Cross-sectional Area of Neo-intimal Tissue Coverage
Description: Cross-sectional area in neointimal hyperplasia by Optical Coherence Tomography (OCT) at 1 year following stent placement
Time Frame: 1 year
Population: The numbers for each different endpoint are dependent on the data quality and availability for each endpoint.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Resolute Integrity DES | Xience Xpedition DES
Number analyzed (Participants) | 32 | 35
mm^2 | 1.381 (1.026) | 0.949 (0.767)

2. Secondary Outcome: In Stent: Mean Thickness of Strut Coverage at Follow up
Description: Mean thickness of strut coverage at follow up (In-Stent safety endpoint). Struts have been considered as covered when tissue overlying the struts is >0 μm by optical coherence tomography (OCT)
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Resolute Integrity DES | Xience Xpedition DES
Number analyzed (Participants) | 32 | 35
mm^2 | 0.118 (0.109) | 0.096 (0.09)

3. Secondary Outcome: In-Stent: Degree of Vascular Straightening Post-percutaneous Coronary Intervention (PCI) (In-Stent Mechanistic Endpoint)
Description: post PCI angulation by Angio: In-Stent: Degree of vascular straightening post-percutaneous coronary intervention (PCI) (In-Stent mechanistic endpoint)
Time Frame: Immediately after stent implantation
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | Resolute Integrity DES | Xience Xpedition DES
Number analyzed (Participants) | 42 | 40
Degree | 40 (25) | 36 (33)

4. Secondary Outcome: In Stent: Plaque Prolapse Post-PCI (In-Stent Mechanistic Endpoint)
Description: Plaque will be identified by Optical Coherence Tomography (OCT)- In-Stent: Plaque prolapse post-PCI (In-Stent mechanistic endpoint)
Time Frame: Immediately after stent implantation
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Resolute Integrity DES | Xience Xpedition DES
Number analyzed (Participants) | 39 | 38
mm^2 | 0.12 (0.14) | 0.13 (0.16)

5. Secondary Outcome: In-Stent: Percent Area of Low Wall Shear Stress (WSS)-(In-Stent Mechanistic Endpoint)
Description: The % area of low wall shear stress immediately after stent implantation will be measured by Optical Coherence Tomography (OCT)
Time Frame: Immediately after stent implantation
Population: This outcome required that patients received computational fluid dynamics analysis, unfortunately, this was not possible in all patients.
Measure: Mean (Standard Deviation); unit: percentage of area
Arm/Group | Resolute Integrity DES | Xience Xpedition DES
Number analyzed (Participants) | 41 | 37
percentage of area | 0.9 (0.13) | 0.9 (0.11)

6. Secondary Outcome: Stent Edge -Change in Plaque Area (Efficacy Endpoint) at 5 mm Proximal and Distal to Stent.
Description: Change in plaque area at the stent edges will be calculated from the change in plaque area in the 5 mm proximal and distal segments by intravascular ultrasound (IVUS); calculated as follow-up values minus baseline values
Time Frame: 1 year
Population: The number of participants with images that are of adequate quality for analysis. The number reported corresponds to the actual change in plaque area between baseline and 1 year follow-up
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Resolute Integrity DES | Xience Xpedition DES
Number analyzed (Participants) | 34 | 31
mm^2 | -0.8 (1.7) | -0.5 (2.8)

7. Secondary Outcome: Stent Edge: Degree of Vascular Straightening Post-percutaneous Coronary Intervention (PCI) at the Stent Edges (Stent Edge Mechanistic Endpoint)
Description: Degree of vascular straightening post-percutaneous coronary intervention (PCI) at the stent edges (Stent Edge mechanistic endpoint) will be measured post PCI angulation by Angio
Time Frame: Immediately after stent implantation
Population: This outcome only requires baseline angiograms hence more patients meet this criteria.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Resolute Integrity DES | Xience Xpedition DES
Number analyzed (Participants) | 42 | 40
Degrees | 22 (14) | 21 (14)

8. Secondary Outcome: Stent Edge: Percent Area With Low Wall Shear Stress (WSS) at Stent Edges Post-PCI (Mechanistic Endpoint)
Description: The % area of low wall shear stress in the 5 mm proximal and distal segments immediately after stent implantation will be measured by intravascular ultrasound (IVUS).
Time Frame: Immediately after stent implantation
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of area
Arm/Group | Resolute Integrity DES | Xience Xpedition DES
Number analyzed (Participants) | 41 | 37
percentage of area | 0.6 (0.23) | 0.64 (0.29)

ADVERSE EVENTS:
Time Frame: All patients were followed while in hospital for major adverse events (starting 12-24Hr post-procedure, up to 1- year).
Arm/Group | Resolute Integrity DES | Xience Xpedition DES
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/41
Serious Adverse Events (participants affected / at risk) | 2/45 | 2/41
Other Adverse Events (participants affected / at risk) | 0/45 | 2/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resolute Integrity DES (N=45) | Xience Xpedition DES (N=41)
Recurrent Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Appendectomy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Balloon Fracture (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resolute Integrity DES (N=45) | Xience Xpedition DES (N=41)
Unstable Angina (Cardiac disorders) | 0 (0) | 1 (1)
Target vessel revascularization (Surgical and medical procedures) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/76/NCT02098876/Prot_SAP_000.pdf
  • Informed Consent Form (2015-12-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT02098876/ICF_001.pdf